CLINICAL TRIAL: NCT00653952
Title: A Phase 3, Randomized, Open-Label, Comparative Study of CAELYX Versus Paclitaxel HCl in Patients With Epithelial Ovarian Carcinoma Following Failure of First-Line, Platinum-Based Chemotherapy
Brief Title: CAELYX Versus Paclitaxel HCl in Patients With Epithelial Ovarian Carcinoma Following Failure of First-Line, Platinum-Based Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Sequus Pharmaceuticals (Industry); ALZA (Industry)
Responsible Party: DIRECTOR MEDICAL LEADER, Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004369; DOXIL-CAN-301
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Ovarian Neoplasms
Keywords: Paclitaxel HCl; CAELYX; DOXIL; Ovarian Carcinoma; Doxorubicin HCl
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental)
  Interventions: Drug: CAELYX
- 002 (Active Comparator)
  Interventions: Drug: Paclitaxel HCl

INTERVENTIONS:
Drug: CAELYX — Dose of 50 mg/m2 by i.v. infusion over 1 hour every 28 days for up to 1 year
  Arms: 001
Drug: Paclitaxel HCl — Dose of 175 mg/m2 by i.v. infusion over 3 hours starting on Day 1 of a 21-day cy
  Arms: 002

SUMMARY:
The objective of this study is to compare the efficacy and safety of CAELYX versus Paclitaxel HCl in patients with epithelial ovarian carcinoma following failure of first-line, platinum-based chemotherapy. The primary endpoint is time to progression (TTP) following treatment with either CAELYX or Paclitaxel HCl; the secondary endpoints are response rates, time to response, duration of response,quality of life assessment, and survival following treatment with either CAELYX or Paclitaxel HCl. Up to a total of 438 protocol-eligible patients with epithelial ovarian carcinoma following failure of first-line, platinum-based chemotherapy will be enrolled in order to obtain 350 evaluable patients.

DETAILED DESCRIPTION:
This is a randomized, open-label, comparative study of CAELYX versus Paclitaxel HCl in the treatment of patients with epithelial ovarian carcinoma following failure of first line chemotherapy with a platinum-based regimen. Patients entering the trial will be stratified prospectively for platinum-sensitivity and bulky disease and analyzed retrospectively for prior anthracycline therapy. Protocol-eligible patients, with measurable disease, who have received no more than one prior regimen, which was platinum-based, will be randomized to receive either a one-hour intravenous infusion of CAELYX, 50 mg/m2 every 28 days, or Paclitaxel HCl, 175 mg/m2 as a 3 hour infusion every 21 days. Patients will be treated for up to one year. It is suggested that responding patients receive at least 6 cycles of treatment. Patients with ongoing clinical benefit may continue study drug upon approval of the sponsor as long as it is in the patient's interest and in the absence of severe toxicity. It is suggested that patients exhibiting a complete response (CR) receive 2 subsequent cycles of treatment. Patients exhibiting partial response (PR) may continue to receive study drug as long as therapeutic benefit is being derived but it is suggested that they receive at least 3 subsequent cycles of study drug. Patients will undergo appropriate radiological imaging (x-ray, CT scan, MRI) to document baseline disease, as well as a chest x-ray and an assessment of left ventricular ejection fraction (LVEF) by MUGA scan within 30 days prior to the first dose of study drug. Patients will be followed weekly for hematological toxicities. Radiological imaging will be repeated every 7-8 weeks to assess disease status. Patients who achieve complete or partial response will be reevaluated 4 weeks later to confirm the initial observation of response. All patients will be followed for a minimum of one year for disease progression and survival. LVEF will be assessed by MUGA scan at baseline, when the cumulative anthracycline dose reaches 300 mg/m2 (500 mg/m2 epirubicin), and after every 2 cycles of CAELYX thereafter. Endomyocardial biopsy is recommended for patients who have received > 400 mg/m2 of CAELYX alone or a cumulative anthracycline dose of > 550 mg/m2 (including CAELYX; 900 mg/m2 if epirubicin). [NOTE: This study was initiated on 7-May-1997. Due to poor accrual, the study enrollment was terminated on 31-Aug-1999. Patients were followed until study completion on 12-Apr-2000. During the preparation of the study report (beginning in May 2003), the sites were re-queried for clarification of safety and survival data.]

DOXIL, dose of 50 mg/m2 by i.v. infusion over 1 hour every 28 days for up to 1 year. Paclitaxel, dose of 175 mg/m2 by i.v. infusion over 3 hours starting on Day 1 of a 21-day cycle for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven (i.e., not borderline) epithelial ovarian carcinoma
* Measurable disease
* Recurrence of disease or disease progression indicative of failure of first-line platinum-based chemotherapy
* Disease-free from prior malignancies for >5 years with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Adequate renal creatinine (<2.5 mg/dL (<220 μmol/L)) & liver function (aspartate amino transferase (AST) and alanine amino transferase (ALT) <2 x upper limit of normal, alkaline phosphatase <2.0 x upper limit of normal, except if attributed to tumor, and bilirubin < upper limit of normal)

Exclusion Criteria:

* Pregnant or breast feeding
* Life expectancy of <3 months
* Prior radiation therapy to more than one-third of hematopoietic sites within 30 days prior to first dose of study drug
* Prior therapy with DOXIL or paclitaxel
* Prior chemotherapy within 28 days of first dose of study drug (or 42 days if subject has received a nitrosourea or mitomycin)
* Treated with high dose therapy supported by bone marrow or peripheral stem cell transplantation at any time

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 1997-05; Study Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate noninferiority with respect to time to progression (TTP) for CAELYX/DOXIL treatment when compared to paclitaxel treatment. | 8 week intervals

SECONDARY OUTCOMES:
Response rates, time to response, duration of response,quality of life assessment, and survival following treatment with either CAELYX or Paclitaxel HCl. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.